CLINICAL TRIAL: NCT06613854
Title: Effect of Early Combination Antihyperglycemic Treatment With Metformin and Oral Semaglutide vs. Metformin and Empagliflozin on Glycemic and Metabolic Control in Individuals With Short Duration Type 2 Diabetes
Brief Title: Effect of Early Combination Antihyperglycemic Treatment on Metabolic Control in Individuals With Type 2 Diabetes
Acronym: E-SEMPA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-SEMPA; 0120-70/2024-2711-3 (Other: National Medical Ethics Committee of the Republic of Slovenia)
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: E-SEMPA; Early Combination Antihyperglycemic Treatment; Metformin; Semaglutide; Empagliflozin; Glycemic Control; Metabolic Control; Type 2 Diabetes; Insulin Resistance; Time in Range; CGM; Continuous Glucose Monitoring; UMC Ljubljana
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — semaglutide; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Semaglutide Arm (Active Comparator): Participants will receive oral semaglutide in addition to metformin (in a steady daily dose of ≥1500 mg), starting with an initial dose of 3 mg. The dose of semaglutide will be increased to 7 mg after 30 days, and then to a maintenance dose of 14 mg once daily after another 30 days that will be continued to week 26. In the case of inadequately controlled glycemia (HbA1c >8.0 % or symptomatic hyperglycemia), rescue treatment with gliclazide will be initiated.
  Interventions: Drug: Oral semaglutide
- Empagliflozin Arm (Active Comparator): Participants will receive oral empagliflozin in a once daily dose of 10 mg in addition to metformin (in a steady daily dose of ≥1500 mg). The dose of empagliflozin will not be subsequently changed during the duration of the study. In the case of inadequately controlled glycemia (HbA1c >8.0 % or symptomatic hyperglycemia), rescue treatment with gliclazide will be initiated.
  Interventions: Drug: Empagliflozin 10 mg
- Control Arm (No Intervention): Participants will receive metformin in a steady daily dose of ≥1500 mg. In the case of inadequately controlled glycemia (HbA1c >8.0 % or symptomatic hyperglycemia), rescue treatment with gliclazide will be initiated.

INTERVENTIONS:
Drug: Oral semaglutide — Semaglutide Oral Tablets will be introduced to the Oral Semaglutide Arm as per protocol for regular therapy introduction.
  Other Names: Rybelsus
  Arms: Oral Semaglutide Arm
Drug: Empagliflozin 10 mg — Empagliflozin Oral Tablets will be introduced to the Empagliflozin Arm as per protocol for regular therapy introduction.
  Other Names: Jardiance
  Arms: Empagliflozin Arm

SUMMARY:
The goal of this clinical trial is to learn if early combination with two antidiabetic drugs further improves blood glucose control compared to a single drug regimen in adults with short duration of type 2 diabetes. It will also learn about the effect of the combination treatment on body weight, body composition, blood lipids, oxidative stress, inflammation, metabolic control, insulin resistance and insulin secretion from pancreas, together with its safety profile. The main questions it aims to answer are:

* Does early combination with two antidiabetic drugs improve blood glucose levels, determined by continuous glucose monitoring system?
* Is early combination treatment as safe as treatment with a single antidiabetic drug?
* Does early combination treatment reduces the need for rescue therapy?
* Does early combination treatment reduces body weight and improves body composition?
* Does early combination treatment improves blood lipid parameters, oxidative stress and inflammation?
* Does early combination treatment improves metabolic parameters?
* Does early combination treatment improves insulin resistance and insulin secretion?

Researchers will compare early combination treatment with metformin and either peroral semaglutide or empagliflozin to a single drug regimen with only metformin to see if the combination treatment works to treat type 2 diabetes.

Participants will:

* Take the combination of two antidiabetic drugs or only metformin for every day for 26 weeks.
* Visit the clinic four times during the study duration for checkups and tests.
* Carry a continuous glucose monitoring sensor for 14 days prior to study visits.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a progressive chronic disease and represents a significant risk factor for morbidity and mortality due to cardiovascular disease. In addition to managing glycemia, the use of antihyperglycemic medications with further and independent cardiovascular benefits is recommended in managing individuals with T2D. These medications primarily include sodium-glucose cotransporter 2 inhibitors (SGLT2i) and glucagon-like peptide-1 receptor agonists (GLP-1RA). Traditionally, treatment of T2D followed a stepwise intensification by adding antihyperglycemic drugs if optimal glycemic control was not achieved. However, current American Diabetes Association guidelines recommend considering early combination therapy at treatment initiation, particularly at high baseline glycated hemoglobin (HbA1c) levels, to shorten the time to achieve glycemic goals.

In everyday clinical practice, however, treatment intensification is often delayed due to clinical inertia, even when glycemic control is suboptimal. Early intensive treatment of T2D has been shown to improve glycemic control, reduce mortality, and lower the risk of both microvascular and macrovascular complications, while also improving the durability of the glycemic effect.

Previous randomized clinical trials on early combination therapy for T2D have primarily focused on glycemic control, as determined by traditional glycemic parameters such as fasting glucose and HbA1c. However, new insights suggest that these measures alone are insufficient for a holistic assessment of glycemic control in diabetes. There is now a recognized need to consider additional indicators of glycemic control, obtained through continuous glucose monitoring (CGM) systems. Furthermore, data are lacking on the direct comparison of the early combination treatment with either SGLT2i or GLP-1RA on top of metformin.

In this 26-week, prospective, open-label, interventional, randomized, single-center clinical trial with a 3-week run-in period, we aim to investigate the effect of early combination treatment with metformin and GLP-1RA or SGLT2i compared to standard monotherapy with metformin and subsequent escalation of antihyperglycemic treatment on glycemic control, as assessed by continuous glucose monitoring systems and HbA1c, body weight, body composition, lipid profile, oxidative stress, inflammation, metabolic control, insulin resistance, and pancreatic beta-cell function in adults with short duration T2D. The primary outcome of the study will be glycemic control, assessed by time in range (TIR).

The study will include individuals of both sexes, of any race or ethnicity, aged between 18 and 70, with a duration of T2D of less than 2 years, HbA1c levels ≤8.0%, on monotherapy with metformin, and naive to treatment with GLP-1RA and SGLT2i.

After the initial 3-week run-in period, patients will be randomized (based on sex, age, and TIR during the run-in period) into three intervention groups in a 1:1:1 ratio:

(i) a control group, continuing metformin monotherapy; (ii) the first study group, receiving metformin and oral semaglutide; and (iii) the second study group, receiving metformin and empagliflozin.

Patients will then be monitored approximately every 13 weeks (3 months) up to 26 weeks (6 months). Prior to randomization, participants will receive a study package containing 3 sensors and 1 reader of the CGM system. The first sensor will be placed on the participants at the start of the run-in period, and subsequent sensors will be self-applied by participants at least 14 days before the last two study visits (at week 13 and week 26).

At each study visit, a review of medical records, a clinical examination, and blood collection for laboratory tests will be conducted. At randomization (week 0) and during the final study visit (week 26), all participants will undergo a modified oral glucose tolerance test (mOGTT) to assess insulin resistance and pancreatic beta-cell function. Additionally, the first 20 participants from each intervention group will undergo whole-body imaging to evaluate body composition. In the case of inadequately controlled glycemia, rescue treatment with gliclazide from the sulfonylurea class will be initiated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for up to 2 years (prior to randomization);
* Aged between 18 and 70 years, both sexes, of any race or ethnicity;
* HbA1c ≤8.0% at randomization;
* Baseline treatment with metformin at a steady daily dose of ≥1500 mg;
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Treatment at any time in the past with SGLT2i, GLP-1RA, or DPP-4 inhibitors;
* Insulin treatment for longer than 2 weeks in the past;
* Body Mass Index below 22 kg/m2 or BMI above 40 kg/m2;
* Chronic kidney disease stages 3-5 (eGFR below 60 ml/min or the presence of albuminuria (urine albumin-to-creatinine ratio above 34 g/mmol);
* Known cardiovascular disease (angina pectoris, history of myocardial infarction, ischemic heart disease, heart failure, known carotid atherosclerosis, objectively proven peripheral arterial disease, or other known atherosclerotic disease at other locations);
* Moderate or severe liver disease (Child-Pugh stage B or C);
* Personal history of pancreatitis;
* Advanced heart failure (NYHA III-IV);
* Retinopathy or maculopathy or their active treatment;
* Pregnancy, expected pregnancy, or breastfeeding;
* Presence of active malignancy or personal history of malignancy within 5 years of study enrollment;
* Personal history of thyroid cancer; personal or family history of multiple endocrine neoplasia type 2 or family history of medullary thyroid carcinoma;
* Chronic inflammatory bowel disease;
* History of bariatric surgery or other gastrointestinal surgery that could affect drug or nutrient absorption;
* Frequent or severe urinary tract infections;
* Presence of a urinary catheter;
* Troublesome and recurrent genital fungal infections;
* Personal history of ketoacidosis;
* Symptomatic hypotension or predisposition to hypovolemia;
* History of organ transplantation;
* Allergy to any component in the semaglutide or empagliflozin oral tablet;
* Any medical or social circumstance that may limit participation in the study (e.g., inability to attend regular study visits);
* Any other condition that, in the opinion of the principal and responsible investigators, may affect the safety or efficacy of the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) | Period of 14 days prior to last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is in the range of 3.9-10.0 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).

SECONDARY OUTCOMES:
Absolute Change in Time in Range (TIR) | Baseline (week 0) and last study visit (week 26)
  Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Absolute Change in Glycated hemoglobin (HbA1c) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in %)
Time above Range (TAR) | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is above 10.0 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Time below Range (TBR) | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is below 3.9 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Time above Range (TAR) - Level 1 Hyperglycemia | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is in the range of 10.1-13.9 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Time above Range (TAR) - Level 2 Hyperglycemia | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is above 13.9 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Time below Range (TBR) - Level 1 Hypoglycemia | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is in the range of 3.0-3.8 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Time below Range (TBR) - Level 2 Hypoglycemia | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is below 3.0 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Time in Tight Range (TITR) | Last study visit (week 26)
  Defined as the time (or percentage of measurements) when the glucose value in the interstitial fluid is in the range of 3.9-7.8 mmol/L. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Coefficient of variation (CV) | Last study visit (week 26)
  A measure of dynamic glucose variability. Calculated as a ratio of glucose concentration standard deviation and mean glucose concentration, expressed as a percentage. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in %).
Mean Time in Range (TIR) | Study visit at week 13 and week 26
  Mean Time in Range (TIR) at study visit at week 13 and week 26. Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in % or in hours and minutes).
Mean glucose concentration | Last study visit (week 26)
  Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in mmol/L).
Proportion of participants with Coefficient of variation (CV) below or equal to 36% | Last study visit (week 26)
  Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in %).
Standard deviation of mean glucose concentration | Last study visit (week 26)
  Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in mmol/L).
Proportion of participants with Time in Range (TIR) above 70% | Last study visit (week 26)
  Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in %).
Proportion of participants with Time in Range (TIR) above 90% | Last study visit (week 26)
  Assesment by Continuous Glucose Monitoring system FreeStyle Libre 2 (in %).
Proportion of participants with Glycated hemoglobin (HbA1c) below 6.5% | Last study visit (week 26)
  Assessment by biochemical methods (in %)
Proportion of participants with Glycated hemoglobin (HbA1c) below 5.7% | Last study visit (week 26)
  Assessment by biochemical methods (in %).
Proportion of participants requiring rescue therapy with gliclazide | Baseline (week 0) to last study visit (week 26)
  Measured in %.
Proportion of participants with severe hypoglycemia | Baseline (week 0) to last study visit (week 26)
  Severe hypoglycemia is an epizode of hypoglycemia requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions. Measured in %.
Proportion of participants with severe adverse events | Baseline (week 0) to last study visit (week 26)
  Severe adverse event is defined as symptoms that significantly affects daily activities. Assessment by patients themselves. Measured in %.
Proportion of patients withdrawing from the trial due to adverse events of the interventional drugs | Baseline (week 0) to last study visit (week 26)
  Assessment by patients themselves. Measured in %.

OTHER OUTCOMES:
Change in Body Weight | Baseline (week 0) and last study visit (week 26)
  Measured in kg.
Proportion of participants with a reduction of Body Weight above or equal to 5% | Baseline (week 0) and last study visit (week 26)
  Measured in %.
Proportion of participants with a reduction of Body Weight above or equal to 10% | Baseline (week 0) and last study visit (week 26)
  Measured in %.
Change in Waist Circumference | Baseline (week 0) and last study visit (week 26)
  Measured in cm.
Change in Visceral Adipose Tissue Mass | Baseline (week 0) and last study visit (week 26)
  Assessment by Dual x-ray absorptiometry. Measured in g.
Change in the Proportion of the Total Body Fat Mass | Baseline (week 0) and last study visit (week 26)
  Assessment by Dual x-ray absorptiometry. Measured in %.
Change in Concentration of Total Cholesterol (TC) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in mmol/L).
Change in Concentration of High Density Lipoprotein Cholesterol (HDL-C) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in mmol/L).
Change in Concentration of Low Density Lipoprotein Cholesterol (LDL-C) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in mmol/L).
Change in Concentration of Triglycerides (TG) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in mmol/L).
Change in Concentration of Apolipoprotein A1 (ApoA1) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in mmol/L).
Change in Concentration of Apolipoprotein B (ApoB) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods (in mmol/L).
Change in Total Antioxidant Status | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Glutathione Peroxidase Activity in Erythrocytes | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Superoxide Dismutase Activity in Erythrocytes | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of Uric Acid | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of Advanced Oxidation Protein Products (AOPP) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of Advanced Glycosylation End Products (AGE) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of 8-Isoprostane | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of high-sensitivity C-reactive protein (hs-CRP) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of Interleukin-6 (IL-6) | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of Beta-hydroxybutyrate | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change in Concentration of Free Fatty Acids | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods.
Change of Insulin Resistance - Matsuda Index | Baseline (week 0) and last study visit (week 26)
  Insulin Resistance will be estimated from Matsuda Index from modified Oral Glucose Tolerance Test (mOGTT). Lower values of Matsuda Index mean a higher level of insulin resistance.
Change of Insulin Resistance - HOMA-IR | Baseline (week 0) and last study visit (week 26)
  Insulin Resistance will be estimated from Homeostasis Model Assessment for Insulin Resistance (HOMA-IR). Higher values of HOMA-IR mean higher insulin resistance.
Change of Insulin Sensitivity - HOMA2-%S | Baseline (week 0) and last study visit (week 26)
  Homeostatic model assessment (HOMA) will be used to calculate insulin sensitivity. It will be reported as HOMA2-%S (where 100% means normal insulin sensitivity). HOMA2-%S is reciprocal of Homeostasis Model Assessment for Insulin Resistance - HOMA-IR.
  Calculated using HOMA2 Calculator v2.2.4, Oxford Centre for Diabetes, Endocrinology and Metabolism; Oxford University, United Kingdom.
Change of Pancreatic Beta Cell Function - HOMA2-%B | Baseline (week 0) and last study visit (week 26)
  Pancreatic Beta Cell Function will be estimated from Homeostasis Model Assessment 2 of B-cell Function (HOMA2-%B), where 100% means normal Beta cell function.
  Calculated with HOMA2 Calculator v2.2.4, Oxford Centre for Diabetes, Endocrinology and Metabolism; Oxford University, United Kingdom.
Change in Concentration of Alanine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Leucine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Isoleucine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Valine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Phenylalanine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Methionine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Lysine | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Glutamate | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Acylcarnitine C5 | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Acylcarnitine C8:1 | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Acylcarnitine C5-OH | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Acylcarnitine C4-OH | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.
Change in Concentration of Acylcarnitine C4-DC | Baseline (week 0) and last study visit (week 26)
  Assessment by biochemical methods, including tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Diabetes Outpatient Clinic, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No